CLINICAL TRIAL: NCT02116725
Title: Effects of Shower Gel With Zinc on Epidermal Regeneration
Brief Title: Zinc Gel and Epidermal Regeneration in Healthy Human Volunteers
Acronym: ZINGEL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Lars Nannestad Jorgensen, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERS-2013-01-LDT
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Denuded Epidermis
MeSH Terms: interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Shower gel with zinc (Experimental): Zinc gel is applied daily (50 µl/cm2) to wound and surrounding noninjured skin.
  Interventions: Other: Shower gel with zinc
- Plain shower gel (Placebo Comparator): Plain shower gel is applied daily (50 µl/cm2) to wound and surrounding noninjured skin.
  Interventions: Other: Plain shower gel
- Distilled water (Sham Comparator): Distilled Water is applied daily (50 µl/cm2) to wound and surrounding noninjured skin.
  Interventions: Other: Distilled water

INTERVENTIONS:
Other: Shower gel with zinc — Standard shower gel (Sanex) supplemented with zinc sulfate.
  Arms: Shower gel with zinc
Other: Plain shower gel — Standard shower gel (Sanex).
  Arms: Plain shower gel
Other: Distilled water — Sterile distilled Water.
  Arms: Distilled water

SUMMARY:
Zinc is an important metal for the maintenance of healthy skin and wound healing. Washing with detergents e.g. shower gels may deplete the zinc stores in the skin.

The purpose of our study is to see whether repeated washing with zinc containing shower gel of superficial wounds will result in increased healing.

DETAILED DESCRIPTION:
Zinc is a trace element abundantly present in skin with a concentration gradient from the upper stratum corneum layer to the basal layer. This fact probably reflects the necessity for zinc as co-factor in numerous enzymes involved in skin homeostasis and wound healing. Theoretically, showering with surfactants increases the loss of zinc by the shedding of the zinc-rich corneocytes. Thus there is a concern that this forced exfoliation will result in suboptimal zinc levels for the maintenance of physiological processes involved in epidermal homeostasis and repair. A logical development would thus be to supplement shower gel with zinc to compensate for this loss.

In 30 healthy volunteers one epidermal wound (10 mm in diameter) is induced by suction and heat on each buttock. The wounds are washed with shower gel containing zinc, placebo shower gel or water (reference). The treatments are allocated by randomization ensuring that 20 wounds are washed with shower gel containing zinc, 20 wounds are washed with placebo shower gel and 20 wounds are washed with water.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* Age between18 and 65 years
* Written informed consent

Exclusion Criteria:

* Smoker
* Active skin disease in test areas
* Hypersensitivity to zinc or any of the shower gel ingredients
* Immunosuppressive treatment
* Pregnant or breastfeeding females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Epidermal regeneration | Day 4
  Epidermal regeneration will be assessed blindly by histomorphometry in hematoxylin-eosin-stained paraffin sections of the wounds and by optical coherence tomography.

SECONDARY OUTCOMES:
Bacterial growth | Day 4
  Swabs are taken from wounds and adjacent, treated skin.
Skin barrier function | Day 4
  Skin barrier function is measured by transepidermal water loss by an instrument from Cortex.
Keratinocyte proliferation | Day 4
  Immunohistochemical detection of Ki67 in paraffin sections of the wounds using mouse monoclonal antibody (MIB-1).
Matrix metalloproteinase (MMP)-1 expression | Day 4
  Immunohistochemical detection of MMP-1 in paraffin sections of the wounds using mouse monoclonal antibody.
Pain | Days 0, 1, 2, 3 and 4
  Pain is assessed on a VAS scale (0-100 mm) by the participant.

OTHER OUTCOMES:
Serum zinc | Day 0
Zinc deposition onto skin | Day 4
  Stratum corneum will be removed by adhesive tape (tape-stripping) for zinc analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Disease Center and Copenhagen Wound Healing Center, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Background] Lansdown AB, Mirastschijski U, Stubbs N, Scanlon E, Agren MS. Zinc in wound healing: theoretical, experimental, and clinical aspects. Wound Repair Regen. 2007 Jan-Feb;15(1):2-16. doi: 10.1111/j.1524-475X.2006.00179.x. PMID 17244314
- [Background] Woodley DT, Kim YH. A double-blind comparison of adhesive bandages with the use of uniform suction blister wounds. Arch Dermatol. 1992 Oct;128(10):1354-7. PMID 1417023
- [Background] Agren MS, Mirastschijski U, Karlsmark T, Saarialho-Kere UK. Topical synthetic inhibitor of matrix metalloproteinases delays epidermal regeneration of human wounds. Exp Dermatol. 2001 Oct;10(5):337-48. doi: 10.1034/j.1600-0625.2001.100506.x. PMID 11589731
- [Background] Malminen M, Koivukangas V, Peltonen J, Karvonen SL, Oikarinen A, Peltonen S. Immunohistological distribution of the tight junction components ZO-1 and occludin in regenerating human epidermis. Br J Dermatol. 2003 Aug;149(2):255-60. doi: 10.1046/j.1365-2133.2003.05438.x. PMID 12932229
- [Background] Agren MS, Chvapil M, Franzen L. Enhancement of re-epithelialization with topical zinc oxide in porcine partial-thickness wounds. J Surg Res. 1991 Feb;50(2):101-5. doi: 10.1016/0022-4804(91)90230-j. PMID 1990212
- [Background] Ferraq Y, Black DR, Theunis J, Mordon S. Superficial wounding model for epidermal barrier repair studies: comparison of Erbium:YAG laser and the suction blister method. Lasers Surg Med. 2012 Sep;44(7):525-32. doi: 10.1002/lsm.22054. Epub 2012 Aug 1. PMID 22865469